CLINICAL TRIAL: NCT04962984
Title: Evaluation of Hypercoagulability by Thrombin Generation Test in Beta-thalassemia Major
Brief Title: Thrombin Generation in Beta-thalassemia Major
Acronym: TG-THAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CPRC 2017/TG THAL-MARTIN/MS
Record Dates: First submitted 2018-09-24; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Beta Thalassemia Major Anemia
Keywords: Beta Thalassemia Major; hypercoagulability; thrombin generation test
MeSH Terms: conditions — beta-Thalassemia; Thrombophilia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- THAL + (Experimental): patients with beta thalassemia major, requiring blood transfusion regimen. Additional blood sampling will be performed before and immediately after transfusion (21 millilters and 24 millilters respectively), on the occasion of 3 programed transfusions (consecutive or not).
  Interventions: Procedure: blood sampling
- THAL - (Sham Comparator): Patients with beta thalassemia trait, matched with THAL + for age and gender. An unique blood sampling of 24 millilters will be performed.
  Interventions: Procedure: blood sampling
- Healthy volunteers (Sham Comparator): healthy subjects, matched with THAL + for age and gender. An unique blood sampling of 24 millilters will be performed.
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — additional blood sampling for coagulation tests

SUMMARY:
This study aims to evaluate the persistence of a hypercoagulable state in chronically-transfused patients with beta thalassemia major, by using the thrombin generation test (performed in whole blood and plasma). Patients will be compared with 2 control groups: 1/ healthy volunteers and 2/ carriers of beta-thalassemia trait

ELIGIBILITY:
Inclusion Criteria:

* Patient with de Beta-thalassemia major
* Patient with regular blood transfusion regimen (every 4 - 6 weeks)
* informed and signed consent
* weight > 30kg
* Hemoglobin > 7g/dL

Exclusion Criteria:

* Emergency situation
* Patients receiving antithrombotic drugs (anticoagulants such as Vitamin K antagonism, heparin or direct oral anticoagulant) or antiplatelet drugs;
* women of childbearing age without contraception
* pregnancy
* deprivation of liberty
* no consent

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of hypercoagulability using endogenous thrombin potential (ETP) between patients and controls | 6 months
  Measurement of the area under the thrombin generation curve (ie ETP) in THAL+ patients, before and after transfusion, as compared with ETP measured in controls groups (THAL- and healthy volunteers)

SECONDARY OUTCOMES:
Evaluation of endogenous thrombin potential's variations before and after transfusion in THAL+ patients over 3 transfusion episodes | 6 months
  Measurement of the area under the thrombin generation curve before and after transfusion in THAL+ patients over 3 transfusion episodes